CLINICAL TRIAL: NCT01474811
Title: HCV-TARGET: Hepatitis C Therapeutic Registry and Research Network - A Longitudinal, Observational Study.
Brief Title: HCV-TARGET- Hepatitis C Therapeutic Registry and Research Network
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1991
Record Dates: First submitted 2011-11-10; First posted 2011-11-18 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis; Hepatitis C; HCV-TARGET; HCV; Observational Study
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All patients will be invited to participate in the HCV-TARGET Biorepository Specimen Bank (BSB).
  The following will be collected: Blood (Serum and DNA).
  All samples will be collected on a voluntary basis and participation in this project will not affect participation in the main study.
  Samples collected will be stored at the University of Florida for up to 15 years after the end of the study (database closure) at which time they will be destroyed. The implementation and use of the BSB specimens is governed by the University of Florida Biospecimen Repository policy to ensure the appropriate use of the deposited samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of the HCV-TARGET study is to establish a nationwide registry of patients undergoing treatment with antiviral therapies for chronic hepatitis C (HCV) at both academic and community practices.

DETAILED DESCRIPTION:
HCV-TARGET is a longitudinal, observational study that will create a carefully maintained research registry of HCV patients treated with antiviral therapies designed to rapidly inform strategies for better management of populations underrepresented in clinical trials, identify and remediate educational gaps relative to treatment guidelines and adverse event management in order to optimize rates of sustained virological response (SVR), and serve as the core resource for important collaborative translational studies utilizing biospecimens and clinical data from diverse patient populations.

HCV-TARGET is a cooperative academic consortium of principal investigators from Clinical and Translational Award (CTSA)-funded academic institutions and community-based sites affiliated with the academic sites in geographic proximity. The Clinical Coordinating Center (CCC) resides at the University of Florida and the Data Coordinating Center (DCC) resides at the University of North Carolina at Chapel Hill.

The HCV-TARGET registry will characterize the population of chronic hepatitis C (HCV) patients who are being treated with antiviral therapies at academic and community sites. Patient characteristics such as age, race, ethnicity, comorbidity, and disease and treatment status will be examined.

HCV-TARGET will also:

1. Provide baseline and treatment response data that will be used to pre-identify candidates for enrollment in future clinical trials. HCV-TARGET will also develop a well-characterized cohort of protease inhibitor treatment failures to be considered for future trials.
2. Establish and maintain data, a specimen bank and other resources for ancillary studies of the pathogenesis, diagnosis, natural history and treatment of HCV infection.

This study will investigate various aspects of treatment response to regimens containing direct-acting antiviral agents for the treatment of chronic hepatitis C, including the following:

* Patients underrepresented in clinical trials of approved antiviral therapies(including African-Americans, patients with cirrhosis, and patients that are considered null responders to treatment.)
* Treatment persistence
* Virological breakthrough
* Impact of viral load measurement on treatment efficacy
* Adverse Event Management and Surveillance.

The secondary aims for this study will investigate the following:

* Sustained virological response (SVR) rates and safety in special populations.
* Surveillance of drug-drug interactions.
* Treatment and management adherence.
* Pretreatment Education in HCV patient population.
* Use of specialty pharmacy for hepatitis C therapy.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age 18 or older) being treated with antiviral HCV treatment regimens that contain telaprevir or boceprevir.

Exclusion Criteria:

* Inability to provide written informed consent.
* Currently participating in another clinical trial of hepatitis C therapeutics. Studies comparing HCV RNA assays are not considered exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult patients: Aged 18 and older with chronic HCV treated with triple therapy (including protease inhibitors).
Sampling Method: Non-Probability Sample
Enrollment: 13559 (Actual)
Dates: Start 2011-11; Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 24 months
  The primary outcome measure is the occurence (yes or no) of SVR, defined as undetectable HCV RNA in serum at least 3 months after stopping therapy. Point estimates and confidence intervals will be calculated to describe the frequency of SVR in various sub-populations enrolled in HCV-TARGET.

SECONDARY OUTCOMES:
Treatment persistence | 24 months
  Treatment persistence will be the duration of treatment measured from the first dose of medication until treatment is discontinued. Reasons for premature discontinuation of treatment will be recorded.
Virological breakthrough | 24 months
  The occurrence of virological breakthrough defined as an increase of HCV RNA by at least 1-log over nadir or to >100 IU if previously undetectable.
Management of adverse events | 24 months
  Specific interventions to manage selected adverse events, such as anemia and skin rash, will be tabulated and described

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Fried, M.D., Principal Investigator — University of North Carolina, Chapel Hill; David R. Nelson, M.D., Principal Investigator — University of Florida
Locations (60):
- United States (55):
  - Mayo Clinic AZ, Phoenix, Arizona
  - Liver Wellness Center, Little Rock, Arkansas
  - Scripps, La Jolla, California
  - UCSD Medical Center, San Diego, California
  - UCSF/San Fran General Hospital, San Francisco, California
  - Univ of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Denver, Colorado
  - Yale University Digestive Diseases, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Atlanta Medical Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Lake Shore Gastroenterology & Liver Disease Inst., Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - John Hopkins University, Lutherville, Maryland
  - Massachussets General Hospital, Boston, Massachusetts
  - Harvard University/ Beth Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Gastro, Minneapolis, Minnesota
  - University Of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi, Oxford, Mississippi
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Ctr, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Southwest CARE Center, Santa Fe, New Mexico
  - Hudson River Healthcare, Beacon, New York
  - North Shore Hospital, Manhasset, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mountain View Medical Center, Valatie, New York
  - Asheville Gastroenterology Assoc, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - Trial Management Associates (TMA), Wilmington, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Austin Hepatitis Center, Austin, Texas
  - MetaClin Research, Inc, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Research Specialist of Texas, Houston, Texas
  - Metropolitan Liver Diseases and Gastroenterology, Annandale, Virginia
  - Bon Secours St. Mary 's Hospital of Richmond (Liver Institute of Virginia), Richmond, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Liver Clinic, Toronto Western Hospital, UHN, Toronto, Ontario, Canada
- Germany (3):
  - RWTH University Hospital, Aachen
  - J. W. Goethe University Hospital, Frankfurt
  - Hanover Medical School, Hanover
- Fundacion de investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Verna EC, Morelli G, Terrault NA, Lok AS, Lim JK, Di Bisceglie AM, Zeuzem S, Landis CS, Kwo P, Hassan M, Manns MP, Vainorius M, Akushevich L, Nelson DR, Fried MW, Reddy KR. DAA therapy and long-term hepatic function in advanced/decompensated cirrhosis: Real-world experience from HCV-TARGET cohort. J Hepatol. 2020 Sep;73(3):540-548. doi: 10.1016/j.jhep.2020.03.031. Epub 2020 Mar 31. PMID 32243960
- [Derived] Reddy KR, Lim JK, Kuo A, Di Bisceglie AM, Galati JS, Morelli G, Everson GT, Kwo PY, Brown RS Jr, Sulkowski MS, Akuschevich L, Lok AS, Pockros PJ, Vainorius M, Terrault NA, Nelson DR, Fried MW, Manns MP; HCV-TARGET Study Group. All-oral direct-acting antiviral therapy in HCV-advanced liver disease is effective in real-world practice: observations through HCV-TARGET database. Aliment Pharmacol Ther. 2017 Jan;45(1):115-126. doi: 10.1111/apt.13823. Epub 2016 Oct 28. PMID 27790729
- [Derived] Terrault NA, Zeuzem S, Di Bisceglie AM, Lim JK, Pockros PJ, Frazier LM, Kuo A, Lok AS, Shiffman ML, Ben Ari Z, Akushevich L, Vainorius M, Sulkowski MS, Fried MW, Nelson DR; HCV-TARGET Study Group. Effectiveness of Ledipasvir-Sofosbuvir Combination in Patients With Hepatitis C Virus Infection and Factors Associated With Sustained Virologic Response. Gastroenterology. 2016 Dec;151(6):1131-1140.e5. doi: 10.1053/j.gastro.2016.08.004. Epub 2016 Aug 24. PMID 27565882
- [Derived] Welzel TM, Nelson DR, Morelli G, Di Bisceglie A, Reddy RK, Kuo A, Lim JK, Darling J, Pockros P, Galati JS, Frazier LM, Alqahtani S, Sulkowski MS, Vainorius M, Akushevich L, Fried MW, Zeuzem S; HCV-TARGET Study Group. Effectiveness and safety of sofosbuvir plus ribavirin for the treatment of HCV genotype 2 infection: results of the real-world, clinical practice HCV-TARGET study. Gut. 2017 Oct;66(10):1844-1852. doi: 10.1136/gutjnl-2016-311609. Epub 2016 Jul 13. PMID 27418632
- [Derived] Saxena V, Koraishy FM, Sise ME, Lim JK, Schmidt M, Chung RT, Liapakis A, Nelson DR, Fried MW, Terrault NA; HCV-TARGET. Safety and efficacy of sofosbuvir-containing regimens in hepatitis C-infected patients with impaired renal function. Liver Int. 2016 Jun;36(6):807-16. doi: 10.1111/liv.13102. Epub 2016 Mar 24. PMID 26923436
- [Derived] Sulkowski MS, Vargas HE, Di Bisceglie AM, Kuo A, Reddy KR, Lim JK, Morelli G, Darling JM, Feld JJ, Brown RS, Frazier LM, Stewart TG, Fried MW, Nelson DR, Jacobson IM; HCV-TARGET Study Group. Effectiveness of Simeprevir Plus Sofosbuvir, With or Without Ribavirin, in Real-World Patients With HCV Genotype 1 Infection. Gastroenterology. 2016 Feb;150(2):419-29. doi: 10.1053/j.gastro.2015.10.013. Epub 2015 Oct 21. PMID 26497081
- [Derived] Sterling RK, Kuo A, Rustgi VK, Sulkowski MS, Stewart TG, Fenkel JM, El-Genaidi H, Mah'moud MA, Abraham GM, Stewart PW, Akushevich L, Nelson DR, Fried MW, Di Bisceglie AM. Virological outcomes and treatment algorithms utilisation in observational study of patients with chronic hepatitis C treated with boceprevir or telaprevir. Aliment Pharmacol Ther. 2015 Apr;41(7):671-85. doi: 10.1111/apt.13095. Epub 2015 Jan 28. PMID 25627020
- See also: Virological outcomes and treatment algorithms utilisation in observational study of patients with chronic hepatitis C treated with boceprevir or telaprevir. — http://www.ncbi.nlm.nih.gov/pubmed/25627020
- See also: Safety profile of boceprevir and telaprevir in chronic hepatitis C: real world experience from HCV-TARGET. — http://www.ncbi.nlm.nih.gov/pubmed/25218788
- See also: Safety and Efficacy of Sofosbuvir-Containing Regimens in Hepatitis C Infected Patients with Impaired Renal Function. — http://www.ncbi.nlm.nih.gov/pubmed/26923436
- See also: Interferon-free therapy for genotype 1 hepatitis C in liver transplant recipients: Real-world experience from the hepatitis C therapeutic registry and research network. — http://www.ncbi.nlm.nih.gov/pubmed/26519873
- See also: Effectiveness of Simeprevir Plus Sofosbuvir, With or Without Ribavirin, in Real-World Patients With HCV Genotype 1 Infection. — http://www.ncbi.nlm.nih.gov/pubmed/26497081
- See also: Effectiveness of Ledipasvir-Sofosbuvir Combination in Patients With Hepatitis C Virus Infection and Factors Associated of Sustained Virologic Response. — http://www.ncbi.nlm.nih.gov/pubmed/27565882
- See also: Effectiveness and safety of sofosbuvir plus ribavirin for the treatment of HCV genotype 2 infection: results of the real-world, clinical practice HCV-TARGET study. — http://www.ncbi.nlm.nih.gov/pubmed/27418632
- See also: Effectiveness and Safety of Sofosbuvir-Based Regimens for Chronic HCV Genotype 3 Infection: Results of the HCV-TARGET Study. — http://www.ncbi.nlm.nih.gov/pubmed/27325691
- See also: Safety and Effectiveness of Ledipasvir and Sofosbuvir, With or Without Ribavirin, in Treatment-Experienced Patients With Genotype 1 Hepatitis C Virus Infection and Cirrhosis — https://www.ncbi.nlm.nih.gov/pubmed/29306043
- See also: Safety and efficacy of current direct-acting antiviral regimens in kidney and liver transplant recipients with hepatitis C: Results from the HCV-TARGET study — https://www.ncbi.nlm.nih.gov/pubmed/28504842
- See also: All-oral direct-acting antiviral therapy in HCV-advanced liver disease is effective in real-world practice: observations through HCV-TARGET database — https://www.ncbi.nlm.nih.gov/pubmed/27790729
- See also: Public-Private Partnership: Targeting Real-World Data for Hepatitis C Direct-Acting Antivirals. — https://www.ncbi.nlm.nih.gov/pubmed/28757271
- See also: Treatment Status of Hepatocellular Carcinoma Does Not Influence Rates of Sustained Virologic Response: An HCV-TARGET Analysis — https://pubmed.ncbi.nlm.nih.gov/31592494/
- See also: Efficacy of Glecaprevir and Pibrentasvir in Patients With Genotype 1 Hepatitis C Virus Infection With Treatment Failure After NS5A Inhibitor Plus Sofosbuvir Therapy — https://pubmed.ncbi.nlm.nih.gov/31401140/